CLINICAL TRIAL: NCT05128214
Title: Aspirin Thromboprophylaxis After First-line Total Hip and Knee Replacement. Comparison With Baseline Low Molecular Weight Heparin Prophylaxis
Brief Title: Aspirin Thromboprophylaxis After First-line Total Hip and Knee Replacement
Acronym: TBP-ASPIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8299
Record Dates: First submitted 2021-10-14; First posted 2021-11-19 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Hip and Knee Prosthesis Implantation
Keywords: Hip prosthesis implantation; Knee prosthesis implantation; Aspirin thromboprophylaxis; Heparin prophylaxis; Thromboembolic complications; Bleeding complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Annually, more than 100,000 total hip prostheses (THA) and more than 100,000 total knee prostheses (TKA) are implanted for osteoarthritis in France, and these figures are set to increase significantly in the future as in all industrialized countries. . Venous thrombosis is a potentially serious complication after PTH and PTG, justifying various prophylactic measures. In France, aggressive prophylaxis with low molecular weight heparin (LMWH) or direct oral anticoagulants (DOA) was until recently recommended, because this drug is considered to be the most effective, at the cost of a bleeding risk implicitly assumed but often poorly. evaluated. A recent publication suggests that the risk of bleeding is currently greater than the risk of a thromboembolic event.

More recently, foreign or international recommendations have broadened the range of these recommendations, notably by introducing aspirin as a possible prophylactic agent. While this molecule is potentially less effective than LMWHs or ADOs, it could decrease the risk of iatrogenic hemorrhage. The introduction of enhanced recovery procedures after surgery (RAAC) could decrease the risk of thrombosis without modifying the risk of bleeding, and thereby improve the cost-benefit ratio of aspirin, justifying its recent inclusion in the current French recommendations when The operated follows such a protocol.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥ 18 years old);
* Patient operated on for a first-line total hip or knee replacement by the principal investigator;
* Patient not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

- Subject having expressed opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient operated on for a first-line total hip or knee replacement by the principal investigator;
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Study of the postoperative thromboembolic complications after implantation of hip and knee prostheses | Files analysed retrospectively from July 01, 2016 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Pédiatrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France